CLINICAL TRIAL: NCT05068154
Title: Comparing Myovista wavECG to NT Pro-BNP for Heart Failure Referral
Brief Title: Myovista vs NT Pro-BNP Heart Failure Referral Tool
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Great Western Hospitals NHS Foundation Trust (Other)
Collaborators: Royal Cornwall Hospitals Trust (Other); Northern Care Alliance NHS Foundation Trust (Other); North Tees and Hartlepool NHS Foundation Trust (Other); Riverside Medical Center (Other); HeartSciences Inc, USA (Unknown)
Responsible Party: Principal Investigator, Dr Badri Chandrasekaran, Consultant Cardiologist, Director of R&I, Great Western Hospitals NHS Foundation Trust
Other Study IDs: GWH0002
Record Dates: First submitted 2021-09-16; First posted 2021-10-05 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-09

CONDITIONS: Heart Failure
Keywords: Diagnosis; Heart Failure; Primary Care
MeSH Terms: conditions — Heart Failure; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Myovista® WavECG™ — The MyoVista wavECG Device uses wavelet signal processing to extract frequency information from the acquired 12-lead ECG signal which is then analysed using artificial intelligence to provide information relating to left ventricular relaxation abnormalities

SUMMARY:
It is hypothesised that the MyoVista wavECG has the potential to show non inferior sensitivity and specificity compared to the current heart failure pathway screening tools of BNP/NT-proBNP and 12 lead resting ECG, but has the advantage of providing a single, familiar, inexpensive point of care test which provides point of care results and can act as a prescreen, or in circumstances replacement to BNP/NTpro-BNP testing, and eliminate a proportion of the unnecessary testing and echo referrals.

A comparative performance analysis of the modalities will form the basis for the study with subsequent reporting on the financial impact and societal benefits of any potential pathway change.

DETAILED DESCRIPTION:
This is a multi-center, non-interventional, single arm, non-inferiority clinical study of the MyoVista wavECG ability to identify primary care patients for referral to secondary care for diagnosis of heart failure (as defined by BSE (British Society of Echocardiography) guidelines for echo), in direct comparison to BNP/NT-proBNP. The study will be conducted at a maximum of 10 investigational secondary care sites within the United Kingdom, and some/all referring primary care centres for each site. Study subjects presenting at primary care with shortness of breath, risk factors for and/or suspicion of heart failure will be referred to secondary care for 2D transthoracic echocardiogram based on borderline and abnormal BNP/NT-proBNP results as part of the current heart failure pathway as defined by the NICE (National Institute for Health and Care Excellence) guidelines, with the MyoVista wavECG used for the conventional 12 lead ECG reporting and comparison purposes only. MyoVista wavECG results will not be used in the diagnosis of a patient, and/or for the basis of a patient referral to echocardiography for the study duration. In commercial use the MyoVista wavECG will be intended for use in a population of patients being considered for such a referral by providing CWT (Continuous Wavelet Transform) and AI (Artificial Intelligence) derived informatics surrounding an overall summary of left ventricular relaxation abnormalities (High Negative, Negative, Borderline, Positive and Highly Positive). The design of this study will allow for an appropriate evaluation of safety and effectiveness for that population.

The study duration will consist of a single visit for all study subjects, after which the subject's participation in the trial will conclude unless longitudinal study inclusion criteria met and agreed at enrollment (Normal BNP/NT-proBNP, MyoVista wavECG result Negative, Borderline, Positive, Highly Positive).

All study subjects will provide written informed consent for the procedures consistent with the study protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects presenting with shortness of breath and risk factors for and/or suspicion of having early-stage heart failure during initial clinical assessment.
2. Informed Consent - The subject provides written informed consent using an Informed Consent Form that is reviewed and approved by the site's Institutional Review Board (IRB).
3. Sinus rhythm - Conventional ECG results show a sinus rhythm and no other contraindicated rhythm abnormalities (see exclusions below)
4. Age - Subject is ≥18 years of age

Exclusion Criteria:

1. Acute Disease - The subject has current acute coronary syndrome, decompensated heart failure, stroke, or previous history of MI.
2. Prior Cardiac Procedures - The subject has received any prior cardiac interventions or surgical therapeutic procedures relating to cardiac abnormalities: valve replacement, pacemaker implantation, coronary artery bypass grafting (CABG), heart transplant, ablation, coronary stent placement, etc.
3. Rhythm Abnormalities - Conventional ECG results indicating a lack of sinus rhythm and/or automatic heart failure pathway RULE IN rhythms including active atrial fibrillation or atrial flutter, left anterior fascicular block, left and/or right bundle branch block
4. Pregnancy - The subject self declares pregnancy at the time of the study testing
5. Chest deformities - The subject has chest deformities that interfere with accurate measurement of ECG (either conventional or wavECG)
6. Measurement Interference - Subjects with central nervous system or musculoskeletal abnormalities that may interfere with accurate acquisition of ECG and/or echocardiogram measurements.
7. Study Participation - The subject is enrolled in another clinical study that may interfere with MyoVista or echocardiogram measurements. Exceptions to this may be approved prior to enrollment.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject recruitment will include individuals presenting with shortness of breath and with risk factors for and/or suspicion of heart failure, who are to be screened as per the UK National Institute for Care and Clinical Excellence (NIICE) guidelines using a conventional 12 lead resting ECG, BNP/NT-proBNP and referred for echocardiography as part of their standard care.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2022-05-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Non-Inferior Sensitivity (%) and Specificity (%) performance of the MyoVista wavECG compared to BNP/NT-proBNP | 6 months for data collection
  Non-Inferior sensitivity/specificity performance of the MyoVista wavECG to identify patients requiring referral to echo for heart failure diagnosis, compared to the BNP/NT-proBNP measurement
Non-Inferior PPV (%) and NPV (%) performance of the MyoVista wavECG compared to BNP/NT-proBNP | 6 months for data collection
  Non-Inferior PPV/NPV performance of the MyoVista wavECG to identify patients requiring referral to echo for heart failure diagnosis, compared to the BNP/NT-proBNP measurement
Economic analysis of the MyoVista wavECG test compared to BNP/NT-proBNP (£GBP) | 6 months for data collection
  Economic analysis of the MyoVista wavECG as a patient referral to echo tool for heart failure diagnosis compared to BNP/NT-proBNP testing, based on performance improvements (sensitivity and specificity) from MyoVista wavECG. Comparison of referral cost implications of improved risk stratification to include MyoVista waveECG test cost/primary care staff time/cardiology staff time/cost of performing echo vs BNP/NT-proBNP test cost/primary care staff time/cardiology staff time/cost of performing echo

SECONDARY OUTCOMES:
Sensitivity (%) and Specificity (%) performance of MyoVista wavECG to identify patients with systolic dysfunction | 6 months for data collection
  MyoVista wavECG ability to identify patients with left ventricular relaxation abnormalities associated impaired systolic function as defined by reduced ejection fraction (<50%)
PPV (%) and NPV (%) performance of MyoVista wavECG to identify patients with systolic dysfunction | 6 months for data collection
  MyoVista wavECG ability to identify patients with left ventricular relaxation abnormalities associated impaired systolic function as defined by reduced ejection fraction (<50%)

OTHER OUTCOMES:
Sensitivity (%) and Specificity (%) performance of the MyoVista wavECG predictive ability | 24 months from subject enrolment
  Patients who returned a normal BNP/NT-proBNP test will be tracked for future visits to primary/secondary care related to cardiovascular disease for a period of 24 mths, allowing an evaluation of the MyoVista wavECG's ability to predict and identify patients likely to experience future disease onset
PPV (%) and NPV (%) performance of the MyoVista wavECG predictive ability | 24 months from subject enrolment
  Patients who returned a normal BNP/NT-proBNP test will be tracked for future visits to primary/secondary care related to cardiovascular disease for a period of 24 mths, allowing an evaluation of the MyoVista wavECG's ability to predict and identify patients likely to experience future disease onset

CONTACTS AND LOCATIONS:
Locations (1):
- Great Western Hospitals NHS Foundation Trust, Swindon, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided